CLINICAL TRIAL: NCT05890365
Title: Increased Risk of Non-alcoholic Fatty Liver Disease in Low Birth Weight Individuals - Extended Validation.
Brief Title: Increased Risk of Non-alcoholic Fatty Liver Disease in Low Birth Weight Individuals
Status: Recruiting | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other); Lund University (Other)
Responsible Party: Principal Investigator, Charlotte Brøns, Principal investigator, Steno Diabetes Center Copenhagen
Other Study IDs: NAFLD validation
Record Dates: First submitted 2023-03-02; First posted 2023-06-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Low Birth Weight
Keywords: Metabolic disease; Adipose tissue biology; Liver fat; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Diseases; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Abdominal subcutaneous adipose tissue biopsies are retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The investigators recently demonstrated a increase in liver fat in early middle-aged LBW compared to normal birth weight (NBW) men, and 20% of the LBW - but none of the normal birth weight (NBW) - men had previously unknown non-alcoholic fatty liver disease (NAFLD). Here the investigators will further examine the Increased risk of non-alcoholic fatty liver disease in low birth weight individuals by performing a validation study.

DETAILED DESCRIPTION:
An adverse fetal environment characterized by low birth weight (LBW) plays a key role in the development of type 2 diabetes (T2D). The investigators recently demonstrated a 3-fold increase in liver fat in 26 early middle-aged LBW compared to 22 normal birth weight (NBW) men, and 20% of the LBW - but none of the normal birth weight (NBW) - men had previously unknown non-alcoholic fatty liver disease (NAFLD). The investigators hypothesize that ectopic fat deposition and NAFLD is among the earliest disease manifestations and on the critical path to the development of more severe cardiometabolic disease in LBW. Here we aim to perform an extended nested case-control screening study to evaluate hepatic steatosis (NAFLD) and fibrosis in early middle-aged, non-obese LBW men and women and NBW controls. In total, 250 LBW men and women (birth weight (BW) <10% of the population) and 50 NBW controls (BW between 50-90% of the population) born at term (weeks 39-41), 35-40 years-of-age will be recruited from the National Danish Birth Registry for the nested case-control NAFLD screening study. The nested case-control NAFLD screening study will serve as a recruitment platform for a subsequent intervention study.

ELIGIBILITY:
Inclusion Criteria:

* 250 healthy, men and women born with a low birth weight (birth weight (BW) <10% of the population) and 50 born with a normal birth weight controls (BW between 50-90% of the population)
* born at term (weeks 39-41)

Exclusion Criteria:

* BMI>35 kg/m2
* Disease/medication known to affect primary outcome
* Self-reported high physical activity level
* Alcohol intake above general recommendations.
* Metabolic/liver disease
* Weight gain/loss of >3 kg within the past 6 months

Ages: 35 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy men and women aged between 35-40 years born with a low (cases) and normal (controls) birth weight. All individuals have to be born at term in either the Copenhagen or Aarhus area.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Liver fat content | 0 minutes
  Liver elastography (FibroScan) and validation by MRS

SECONDARY OUTCOMES:
Liver fibrosis | 0 minutes
  Liver elastography, validation by MR and liver histology
Body composition | 0 minutes
  DEXA
Fasting glucose | 0 minutes
  mmol/l
Fasting insulin/C-peptide | 0 minutes
  pmol/l
Fasting lipids | 0 minutes
  mmol/l
Fasting liver enzymes | 0 minutes
  U/L

OTHER OUTCOMES:
Transcriptomics in SAT and ex vivo cultured preadipocytes | 0 minutes
  RNAseq
Epigenetics of SAT and ex vivo cultured preadipocytes | 0 minutes
  Genome-wide DNA methylation
Functional characterization of lipid accumulation | 0 minutes
  Metabolism of ex vivo differentiated preadipocytes
Functional characterization of lipolysis | 0 minutes
  Metabolism of ex vivo differentiated preadipocytes
Functional characterization of glycolysis | 0 minutes
  Metabolism of ex vivo differentiated preadipocytes
Functional characterization of respiration | 0 minutes
  Metabolism of ex vivo differentiated preadipocytes
Adipocyte size | 0 minutes
  Histology in SAT
Adipocyte collagen content | 0 minutes
  Histology in SAT
Immunohistochemical markers of fibrosis | 0 minutes
  Histology in SAT
Immunohistochemical markers of senescence | 0 minutes
  Histology in SAT
Immunohistochemical markers of inflammation | 0 minutes
  Histology in SAT
Adipokine secretion of differentiating preadipocytes | 0 minutes
  Targeted adipokine analysis using immunoassay-based panels

CONTACTS AND LOCATIONS:
Overall Officials: Allan Vaag, MD, PhD, Study Director — Steno Diabetes Center Copenhagen; Charlotte Brøns, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark